CLINICAL TRIAL: NCT01028716
Title: Nonmyeloablative Hematopoietic Cell Transplantation (HCT) for Patients With Hematologic Malignancies Using Related, HLA-Haploidentical Donors: A Phase II Trial of Peripheral Blood Stem Cells (PBSC) as the Donor Source
Brief Title: Donor Peripheral Blood Stem Cell Transplant in Treating Patients With Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study experienced lower accrual rates after the onset of COVID. Upon review of the collected data it was deemed that an adequate amount of subjects has been enrolled to date to assess study aims.
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Principal Investigator, Rachel Salit, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2372.00; NCI-2009-01433 (Other: CTRP (Clinical Trial Reporting Program)); 2372; 2372.00 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9213052 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Acute Biphenotypic Leukemia; Acute Erythroid Leukemia in Remission; Acute Leukemia in Remission; Acute Lymphoblastic Leukemia in Remission; Acute Myeloid Leukaemia With Prior Myelodysplastic Syndrome; Acute Myeloid Leukemia in Remission; Acute Myeloid Leukemia With FLT3/ITD Mutation; Acute Myeloid Leukemia With Inv(3)(Q21Q26.2); RPN1-EVI1; Acute Myeloid Leukemia With Multilineage Dysplasia; Acute Myeloid Leukemia With t(6;9); Acute Undifferentiated Leukemia; Adult Acute Lymphoblastic Leukemia in Complete Remission; B Acute Lymphoblastic Leukemia With T(1;19)(Q23;P13.3); E2A-PBX1 (TCF3-PBX1); Ph+ ALL; Burkitt Lymphoma; Childhood Acute Lymphoblastic Leukemia in Complete Remission; DS Stage II Plasma Cell Myeloma; DS Stage III Plasma Cell Myeloma; Myelodysplastic Syndrome; Recurrent Anaplastic Large Cell Lymphoma; Blasts Under 5 Percent of Bone Marrow Nucleated Cells; Recurrent Follicular Lymphoma; Recurrent Hodgkin Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma; Secondary Acute Myeloid Leukemia; T Lymphoblastic Lymphoma; Hematopoietic Cell Transplant Recipient
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Burkitt Lymphoma; Myelodysplastic Syndromes; Lymphoma, Large-Cell, Anaplastic; Lymphoma, Follicular; Hodgkin Disease; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Multiple Myeloma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclophosphamide; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation; Tacrolimus; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nonmyeloablative HCT, TBI) (Experimental): Patients receive fludarabine IV over 30-60 minutes daily on days -6 through -2 and cyclophosphamide IV over 1-2 hours on days -6, -5, and 3-4. Patients undergo total-body irradiation on day -1. Patients undergo donor peripheral blood stem cell transplant on day 0. Patients then receive tacrolimus IV once daily or PO BID on days 5-180 (may be continued if active GvHD is present), mycophenolate mofetil IV or PO TID on days 5-35 (may be continued if GvHD present), and filgrastim IV beginning on day 5 until the ANC is >= 1,000/mm^3 for three consecutive days.
  Interventions: Drug: Cyclophosphamide; Biological: Filgrastim; Drug: Fludarabine Phosphate; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Tacrolimus; Radiation: Total-Body Irradiation

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Filgrastim — Given SQ
  Other Names: Filgrastim XM02; Filgrastim-sndz; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim; Zarxio
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplantation — Undergo PBSC
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplantation; NST
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo PBSC
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Drug: Tacrolimus — Given IV or PO
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic
Radiation: Total-Body Irradiation — Undergo total-body irradiation (TBI)
  Other Names: TOTAL BODY IRRADIATION; Whole-Body Irradiation

SUMMARY:
This phase II trial studies how well donor peripheral blood stem cell (PBSC) transplant works in treating patients with hematologic malignancies. Cyclophosphamide when added to tacrolimus and mycophenolate mofetil is safe and effective in preventing severe graft-versus-host disease (GVHD) in most patients with hematologic malignancies undergoing transplantation of bone marrow from half-matched (haploidentical) donors. This approach has extended the transplant option to patients who do not have matched related or unrelated donors, especially for patients from ethnic minority groups. The graft contains cells of the donor's immune system which potentially can recognize and destroy the patient's cancer cells (graft-versus-tumor effect). Rejection of the donor's cells by the patient's own immune system is prevented by giving low doses of chemotherapy (fludarabine phosphate and cyclophosphamide) and total-body irradiation before transplant. Patients can experience low blood cell counts after transplant. Using stem cells and immune cells collected from the donor's circulating blood may result in quicker recovery of blood counts and may be more effective in treating the patient's disease than using bone marrow.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate that use of PBSC in place of marrow as the source of lymphocytes and stem cells for nonmyeloablative transplants from related, haploidentical donors will not result in unacceptable rates of high-grade acute or chronic GVHD, non-relapse mortality or relapse compared to historical data on nonmyeloablative transplants from unrelated donors.

SECONDARY OBJECTIVES:

I. Estimates of the rates of neutrophil and platelet recovery, number of red blood cell (RBC) and platelet transfusions, incidences of graft failure, transplant-related toxicities, disease-free survival and overall survival.

OUTLINE:

Patients receive fludarabine intravenously (IV) over 30-60 minutes daily on days -6 through -2 and cyclophosphamide IV over 1-2 hours on days -6, -5, and 3-4. Patients undergo total-body irradiation on day -1. Patients undergo donor peripheral blood stem cell transplant on day 0. Patients then receive tacrolimus IV once daily or orally (PO) twice daily (BID) on days 5-180 (may be continued if active GVHD is present), mycophenolate mofetil IV or PO thrice daily (TID) on days 5-35 (may be continued if GVHD present), and filgrastim IV beginning on day 5 until the absolute neutrophil count (ANC) is >= 1,000/mm^3 for three consecutive days.

Treatment continues in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Molecular based human leukocyte antigen (HLA) typing will be performed for the HLA-A, -B, -Cw, -DRB1 and -DQB1 loci to the resolution adequate to establish haplo-identity; a minimum match of 5/10 is required; an unrelated donor search is not required for a patient to be eligible for this protocol if the clinical situation dictates an urgent transplant; clinical urgency is defined as 6-8 weeks from referral or low-likelihood of finding a matched, unrelated donor
* Acute leukemias (includes T lymphoblastic lymphoma); remission is defined as < 5% blasts with no morphological characteristics of acute leukemia (e.g., Auer rods) in a bone marrow with > 20% cellularity, peripheral blood counts showing ANC > 1000/ul, including patients in complete remission with incomplete platelet recovery (CRp); if the marrow has < 20% cellularity due to treatment related cytotoxicity, but still has < 5% blasts, an exception may be made to include this patient up to principal investigator (PI) discretion
* Acute lymphoblastic leukemia in high risk first complete remission (CR1) as defined by at least one of the following:

  * Adverse cytogenetics including but not limited to t(9;22), t(1;19), t(4;11), mixed lineage leukemia (MLL) rearrangements
  * White blood cell counts > 30,000/mcL
  * Patients over 30 years of age
  * Time to complete remission > 4 weeks
  * Presence of extramedullary disease
  * Minimal residual disease
  * Other risk factors determined by the patient's attending physician to be high risk features requiring transplantation
* Acute myelogenous leukemia in high risk CR1 as defined by at least one of the following:

  * Greater than 1 cycle of induction therapy required to achieve remission
  * Preceding myelodysplastic syndrome (MDS)
  * Presence of fms-like tyrosine kinase receptor-3 (Flt3) abnormalities
  * French-American-British (FAB) M6 or M7 leukemia, or
  * Adverse cytogenetics for overall survival such as:

    * Those associated with MDS
    * Complex karyotype (>= 3 abnormalities); or
    * Any of the following: inv(3) or t(3;3), t(6;9), t(6;11), + 8 [alone or with other abnormalities except for t(8;21), t(9;11), inv(16) or t(16;16)], t(11;19)(q23;p13.1)]
  * Other risk factors determined by the patient's attending physician to be high risk features requiring transplantation
* Acute leukemias in second (2nd) or subsequent remission
* Biphenotypic/undifferentiated leukemias in first (1st) or subsequent complete remission (CR)
* High-risk MDS status-post cytotoxic chemotherapy
* Burkitt's lymphoma: second or subsequent CR
* Chemotherapy-sensitive (at least stable disease) large cell, mantle cell or Hodgkin's lymphomas that have failed at least 1 prior regimen of multi-agent chemotherapy and are ineligible for an autologous transplant
* Marginal zone B-cell lymphoma or follicular lymphoma that has progressed after at least two prior therapies (excluding single agent Rituxan)
* Multiple myeloma (MM) stage II or III patients who have progressed after an initial response to chemotherapy or autologous hematopoietic stem cell transplantation (HSCT) or MM patients with refractory disease who may benefit from tandem autologous-nonmyeloablative allogeneic transplant
* Left ventricular ejection fraction at rest must be >= 35%
* Bilirubin =< 2.5 mg/dL
* Alanine aminotransferase (ALT) < 5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) < 5 x ULN
* Alkaline phosphatase < 5 x ULN
* Serum creatinine within normal range for age, or if serum creatinine outside normal range for age, then renal function (creatinine clearance or glomerular filtration rate [GFR]) > 40 mL/min/1.73m^2
* Forced expiratory volume in one second (FEV1), forced vital capacity (FVC), diffusion capacity of carbon monoxide (DLCO) (diffusion capacity) >= 40% predicted (corrected for hemoglobin); if unable to perform pulmonary function tests, then oxygen (O2) saturation > 92% on room air
* Karnofsky/Lansky score >= 60%
* Patients who have received a prior allogeneic HSCT and who have either rejected their grafts or who have become tolerant of their grafts with no active GVHD requiring immunosuppressive therapy
* Patients will undergo standard pre-transplant work-up as dictated by standard practice guidelines the results of which may be used for screening for this study
* DONOR: Donors must be HLA-haploidentical first-degree relatives of the patient; eligible donors include biological parents, siblings, or children, or half-siblings
* DONOR: Age >= 12 years
* DONOR: Weight >= 40 kg
* DONOR: Ability of donors < 18 years of age to undergo apheresis without use of a vascular access device; vein check must be performed and verified by an apheresis nurse prior to arrival at the Seattle Cancer Care Alliance (SCCA)
* DONOR: Donors must meet the selection criteria as defined by the Foundation for the Accreditation of Cell Therapy (FACT) and will be screened per the American Association of Blood Banks (AABB) guidelines

Exclusion Criteria:

* HLA-matched or single allele-mismatched donor able to donate
* Pregnancy or breast-feeding
* Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings)
* Patients with primary idiopathic myelofibrosis
* DONOR: Positive anti-donor HLA antibody

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-05-19 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel B. Salit, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Nonmyeloablative HCT, TBI): Conditioning: Fludarabine IV over 30-60 minutes daily on days -6 through -2 and cyclophosphamide IV over 1-2 hours on days -6, -5, and 3-4. Patients undergo total-body irradiation on day -1.
  Cell product: Patients undergo donor peripheral blood stem cell transplant on day 0.
  GVHD Prophylaxis: Patients then receive tacrolimus IV once daily or PO BID on days 5-180 (may be continued if active GvHD is present), mycophenolate mofetil IV or PO TID on days 5-35 (may be continued if GvHD present), and filgrastim IV beginning on day 5 until the ANC is >= 1,000/mm^3 for three consecutive days.
Period: Overall Study
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Started | 46
Completed | 45
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 45
Age, Continuous [Median (Full Range); unit: years] | 52 [12 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 32
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Non-relapse Mortality at 1 Year
Description: Cumulative incidence of death without evidence of disease progression at 1 year
Time Frame: Up to 1 year
Measure: Number; unit: percent of participants
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 45
percent of participants | 22

2. Primary Outcome: Percentage of Participants With Chronic Graft Versus Host Disease
Description: Scored according to the National Cancer Institute criteria. Mild-to-severe chronic GVHD at 2 years.
Time Frame: Up to 2 years post-transplant
Population: Patients who were alive greater than day 100 were included
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 41
percentage of participants | 26

3. Primary Outcome: Incidence of Grades III/IV Acute Graft Versus Host Disease
Description: Grading determined by organ system stages. Grade III/IV acute graft versus host disease is defined as skin: stage IV, liver: stages II-IV, and/or gastrointestinal tract: stages II-IV.
Time Frame: At day 84
Measure: Number; unit: percent
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 45
percent | 82

4. Primary Outcome: Relapse of Malignancy After Transplantation
Description: Defined by either morphological or cytogenetic evidence of acute leukemia consistent with pre-transplant features, or radiologic evidence of lymphoma progression. When in doubt, the diagnosis of recurrent or progressive lymphoma should be documented by tissue biopsy.
Time Frame: Up to 7 years
Measure: Number; unit: percent
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 45
percent | 29

5. Secondary Outcome: Time to Neutrophil Recovery
Description: Achievement of an absolute neutrophil count greater or equal to 500/mm^3 for three consecutive measurements on different days. The first of the three days will be designated the day of neutrophil recovery.
Time Frame: Up to day 84 post-transplant
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 45
days | 16 [13 to 29]

6. Secondary Outcome: Time to Platelet Recovery
Description: The first day of a sustained platelet count > 20,000/mm^3 with no platelet transfusions in the preceding seven days.
Time Frame: Up to day 84 post-transplant
Measure: Median (Full Range); unit: days
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 42
days | 23 [17 to 50]

7. Secondary Outcome: Incidence of Primary Graft Failure
Description: Defined as < 5% donor CD3 chimerism. Chimerism will be measured by short tandem repeat-polymerase chain reaction on peripheral blood sorted into CD3 and CD33 cell fractions.
Time Frame: At day 84
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 45
Participants | 0

8. Secondary Outcome: Disease-free Survival
Description: Defined as being alive and in remission by < 5% blasts by bone marrow morphology for patients with myeloid malignancies and CT or PET imaging for patients with lymphoid malignancies at the time of the assessment
Time Frame: 3 years from the date of transplant
Measure: Number; unit: percent of participants
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 45
percent of participants | 40

9. Secondary Outcome: Toxicity of Treatment Regimen Determined by Number of Adverse Events Per Organ System
Description: Assessed by Common Terminology Criteria for Adverse Events version 3.0. The incidence of all adverse events greater or equal to grade 3 was determined.
Time Frame: Up to day 90
Measure: Number; unit: events
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 45
events
  Cardiac | 13
  Fever | 9
  Rash | 4
  Gastrointestinal | 17
  Infections | 55
  CMV Reactivation | 26
  Febrile Neutropenia | 25
  Metabolic/laboratory | 24
  Musculoskeletal | 3
  Neurologic | 5
  Pain | 6
  Pulmonary | 10
  Renal/Genitourinary | 10

10. Secondary Outcome: Number of Red Blood Cell Transfusions
Description: Number of units of RBCs given to the patient between day 0 and day 100 post transplant
Time Frame: Day 0-100
Measure: Median (Full Range); unit: transfusions
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 45
transfusions | 8 [0 to 32]

11. Secondary Outcome: Number of Platelet Transfusions
Description: Number platelet transfusions given to the patient between day 0 and day 100 post transplant
Time Frame: Day 0-100
Measure: Median (Full Range); unit: transfusions
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 45
transfusions | 6 [1 to 52]

12. Secondary Outcome: Point Estimate of Overall Survival at 3 Years
Description: Kaplan Meier estimate of the percentage of participants with overall survival at 3 years
Time Frame: 3 years
Measure: Number; unit: percent
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
Number analyzed (Participants) | 45
percent | 45.3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 100 days post HCT. Serious Adverse Events were collected until 1 year post-HCT. All cause mortality was assessed up to 3 years post transplant.
Arm/Group | Treatment (Nonmyeloablative HCT, TBI)
All-Cause Mortality (participants affected / at risk) | 21/45
Serious Adverse Events (participants affected / at risk) | 4/45
Other Adverse Events (participants affected / at risk) | 44/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nonmyeloablative HCT, TBI) (N=45)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (2) — Rehospitalization for acute hypoxemic respiratory failure
Heart Failure (Cardiac disorders) | 1 (1) — Worsening dyspnea with drop in EF to 35%
Diffuse Alveolar Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) — DAH requiring intubation and ICU admission. Resulted in Death.
Acute hypoxemia respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Nonmyeloablative HCT, TBI) (N=45)
Cardiac (Cardiac disorders) | 13 (13) — including arrythmia
Infection (Infections and infestations) | 42 (115) — Including episodes of febrile neutropenia, infections and viral reactivations with BK and CMV in the blood.
Pain (Musculoskeletal and connective tissue disorders) | 6 (9)
Metabolic (Metabolism and nutrition disorders) | 15 (24)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 10 (10)
GI (Gastrointestinal disorders) | 13 (17)
Renal (Renal and urinary disorders) | 5 (10)
Derm (Skin and subcutaneous tissue disorders) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-13): https://cdn.clinicaltrials.gov/large-docs/16/NCT01028716/Prot_SAP_000.pdf